CLINICAL TRIAL: NCT07253688
Title: Adjunctive Rifampin for the Treatment of Prosthetic Valve Endocarditis Due to S. Aureus (RIFA-SNAP)
Brief Title: Adjunctive Rifampin for the Treatment of Prosthetic Valve Endocarditis Due to S. Aureus
Acronym: RIFA-SNAP
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Todd C. Lee MD MPH FIDSA (Other)
Collaborators: McGill University Health Centre/Research Institute of the McGill University Health Centre (Other); Canadian Institutes of Health Research (CIHR) (Other Government); University of Melbourne (Other); The Peter Doherty Institute for Infection and Immunity (Other)
Responsible Party: Sponsor-Investigator, Todd C. Lee MD MPH FIDSA, Professor of Medicine, McGill University Health Centre/Research Institute of the McGill University Health Centre
Organization: McGill University Health Centre/Research Institute of the McGill University Health Centre (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2025-10882
Record Dates: First submitted 2025-11-19; First posted 2025-11-28 (Actual); Last update posted 2025-12-10 (Actual); Status verified 2025-12

CONDITIONS: Staphylococcus Aureus Endocarditis; Prosthetic Valve Endocarditis
Keywords: S. aureus bacteremia; Prosthetic valve endocarditis; Rifampin
MeSH Terms: interventions — Rifampin

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: The trial analyst will also be blinded.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- No rifampin (Experimental): These patients will not receive adjunctive rifampin.
  Interventions: Other: No rifampin
- Adjunctive rifampin (Active Comparator): These patients will receive adjunctive rifampin as recommended in guidelines.
  Interventions: Drug: Rifampin

INTERVENTIONS:
Drug: Rifampin — Patients will receive rifampin 900mg a day in 2-3 divided doses
  Arms: Adjunctive rifampin
Other: No rifampin — Subjects will be assigned to not receive adjunctive rifampin
  Arms: No rifampin

SUMMARY:
This is a sub-study of the S. aureus Network Adaptive Platform (SNAP) trial (NCT05137119) wherein we will evaluate whether not giving rifampin in patients with probable or definite prosthetic valve endocarditis due to S. aureus is non-inferior to giving rifampin.

ELIGIBILITY:
Inclusion Criteria:

1. Probable or definite prosthetic valve endocarditis involving the tricuspid, pulmonic, mitral and/or aortic valves by the 2023 Duke-ISCVID Criteria (including Cardiac PET evidence if applicable);
2. Patient or healthcare proxy provide informed consent.

Exclusion Criteria:

1. Death deemed imminent and inevitable within days or patient will be receiving palliative care and has prognosis < 90 days according to the treating team;
2. Patient requires intensive care but has a do not resuscitate order precluding transfer;
3. Polymicrobial bacteremia (not including skin commensals or other recognized contaminant);
4. Organism tests as rifampin resistant;
5. History of hypersensitivity/anaphylaxis or severe adverse reaction to rifampin;
6. Category X or other important drug-drug interaction with rifampin which cannot be safely mitigated [with as-needed consultation from experts from pharmacy and/or internal medicine/geriatrics for potential deprescribing];
7. Child Pugh Class C cirrhosis;
8. Clinician deems rifampin to be mandatory;
9. Patient has already received >3 days of rifampin at time of screening or >10 days of total therapy
10. Pregnancy or breast feeding

Administrative exclusions:

1. No reliable means of outpatient contact (telephone/email/text);
2. Previously enrolled;
3. Prior S. aureus bacteremia within the preceding 180 days

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 330 (Estimated)
Dates: Start 2025-11-10 (Actual); Primary Completion 2029-12 (Estimated); Study Completion 2030-07 (Estimated)

PRIMARY OUTCOMES:
Treatment failure | 180 days
  A composite outcome of all cause mortality, unplanned cardiac surgery, new cardioembolic events, or relapse of bacteremia due to S. aureus.

SECONDARY OUTCOMES:
All-cause mortality | 180 days
  Death due to any cause
Unplanned cardiac surgery | 180 days
  The need for cardiac surgery which was not planned or scheduled at the time of randomization.
New embolic events | 180 days
  A new symptomatic cardio-embolic event occurring after randomization.
Relapse of bacteremia | 180 days
  A new S. aureus bacteremia with the same susceptibility pattern (except for quinolones or rifampin in those who are exposed) which develops after sterilization of the initial blood cultures
Discontinuation of rifampin due to new drug-drug interaction | 56 days
  The cessation of adjunctive rifampin due to a new pharmacologically significant drug-drug interaction.
Serious adverse drug reaction due to rifampin | 56 days
  Patients who have a CTCAE grade 4 reaction which is determined by expert adjudication to be probably or definitely due to rifampin.
Discontinuation of rifampin due to an adverse drug reaction | 56 days
  Any adverse drug reaction which leads to the discontinuation of rifampin

OTHER OUTCOMES:
Development of rifampin resistant S. aureus | 180 days
  Any clinically relevant isolate of S. aureus which demonstrates resistance to rifampin.

CONTACTS AND LOCATIONS:
Locations (1):
- McGill University Health Centre (Royal Victoria Hospital and Montreal General Hospital), Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: Undecided
Data sharing policies are dependent on the policies of the SNAP Platform (NCT05137119)

REFERENCES:
- [Background] Ryder JH, Tong SYC, Gallagher JC, McDonald EG, Thevarajan I, Lee TC, Cortes-Penfield NW. Deconstructing the Dogma: Systematic Literature Review and Meta-analysis of Adjunctive Gentamicin and Rifampin in Staphylococcal Prosthetic Valve Endocarditis. Open Forum Infect Dis. 2022 Oct 31;9(11):ofac583. doi: 10.1093/ofid/ofac583. eCollection 2022 Nov. PMID 36408468
- [Background] McDonald EG, Aggrey G, Aslan AT, Casias M, Cortes-Penfield N, Dong MQD, Egbert S, Footer B, Isler B, King M, Maximos M, Wuerz TC, Azim AA, Alza-Arcila J, Bai AD, Blyth M, Boyles T, Caceres J, Clark D, Davar K, Denholm JT, Forrest G, Ghanem B, Hagel S, Hanretty A, Hamilton F, Jent P, Kang M, Kludjian G, Lahey T, Lapin J, Lee R, Li T, Mehta D, Moore J, Mowrer C, Ouellet G, Reece R, Ryder JH, Sanctuaire A, Sanders JM, Stoner BJ, So JM, Tessier JF, Tirupathi R, Tong SYC, Wald-Dickler N, Yassin A, Yen C, Spellberg B, Lee TC. Guidelines for Diagnosis and Management of Infective Endocarditis in Adults: A WikiGuidelines Group Consensus Statement. JAMA Netw Open. 2023 Jul 3;6(7):e2326366. doi: 10.1001/jamanetworkopen.2023.26366. PMID 37523190
- See also: Main Website for the S. aureus Network Adaptive Platform Trial (SNAP) — https://www.snaptrial.com.au/